CLINICAL TRIAL: NCT03993327
Title: Pilot Study: Detection of Colorectal Metastatic Liver Disease Preoperatively Using 124I-Labeled M5A Monoclonal Antibody to Carcinoembryonic Antigen (CEA)
Brief Title: An Imaging Agent (I-124 M5A) in Detecting CEA-Positive Liver Metastases in Patients With Colorectal Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 18386; NCI-2019-01923 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 18386 (Other: City of Hope Medical Center)
Record Dates: First submitted 2019-06-04; First posted 2019-06-20 (Actual); Last update posted 2024-06-28 (Actual); Status verified 2024-06

CONDITIONS: Colorectal Carcinoma Metastatic in the Liver; Metastatic Colorectal Carcinoma; Stage IV Colorectal Cancer AJCC v8; Stage IVA Colorectal Cancer AJCC v8; Stage IVB Colorectal Cancer AJCC v8; Stage IVC Colorectal Cancer AJCC v8
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Diagnostic (iodine I 124 monoclonal antibody M5A, PET scan) (Experimental): Patients receive iodine I 124 monoclonal antibody M5A IV on day 0 and undergo PET scan on days 2 and 6.
  Interventions: Biological: Iodine I 124 Monoclonal Antibody M5A; Procedure: Positron Emission Tomography

INTERVENTIONS:
Biological: Iodine I 124 Monoclonal Antibody M5A — Given IV
  Other Names: 124I-M5A; Iodine I 124 Anti-CEA Monoclonal Antibody M5A
Procedure: Positron Emission Tomography — Undergo PET scan
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging

SUMMARY:
This phase I trial studies how well an imaging agent called I-124 M5A works in detecting CEA-positive colorectal cancer that has spread to the liver. I-124 M5A is a monoclonal antibody, called M5A, linked to a radioactive substance called I-124. M5A binds to CEA-positive cancer cells and may, through imaging scans, be able to detect liver metastases by picking up signals from I-124.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the ability of iodine I 124 monoclonal antibody M5A (124I-labeled M5A monoclonal antibody [MAb]) to localize to CEA positive gastrointestinal (GI) metastases primarily focused on the liver.

SECONDARY OBJECTIVES:

I. To determine the safety and pharmacokinetics of administration of 124I-labeled M5A MAb.

II. To correlate the radiographic positron emission tomography (PET) images to the liver metastases pathology.

III. To assess if the I-124 imaging agent detected additional liver and additional extra-hepatic liver lesions not appreciated on standard imaging scans.

OUTLINE:

Patients receive iodine I 124 monoclonal antibody M5A intravenously (IV) on day 0 and undergo PET scan on days 2 and 6.

After completion of study, patients are followed up periodically for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed metastatic colorectal cancer with liver metastases. NOTE: We are not requiring proof of CEA positive disease because > 95% of colorectal cancers are CEA positive
* The effects of 124I-M5A on the developing fetus are unknown. For this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control or abstinence) prior to study entry and for six months following duration of study participation. Should a woman become pregnant or suspect that she is pregnant while participating on the trial, she should inform her treating physician immediately
* Patients must have at least 2 known sites of metastatic liver disease. Patients should have at least one resectable liver metastasis as assessed by hepatobiliary surgical oncology
* The results of the imaging scans that are performed as part of the standard work up should be available and should have been done within 2 months prior to study entry
* All subjects must have the ability to understand and the willingness to sign a written informed consent
* Prior therapy (chemotherapy, immunotherapy, radiotherapy) must be completed at least 2 weeks prior to infusion of radiolabeled antibody

Exclusion Criteria:

* Patients should not have any uncontrolled illness including ongoing or active infection
* Patients who have allergy to iodine or iodine contrast agents are not eligible for this protocol
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to 124I-M5A
* Patients must not have received prior chemotherapy or radiation for >= 2 weeks before study enrollment
* Pregnant women are excluded from this study because 124I-M5A is an agent with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with 124I-M5A, breastfeeding should be discontinued if the mother is treated with 124I-M5A
* Patients with single (= 1) liver metastasis are not eligible for this protocol
* Any patient who has had exposure to mouse, chimeric (human/mouse) or humanized immunoglobulin and has antibody to the M5A
* Subjects, who in the opinion of the investigator, may not be able to comply with the safety monitoring requirements of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2020-07-15 (Actual); Primary Completion 2024-06-04 (Actual); Study Completion 2024-06-04 (Actual)

PRIMARY OUTCOMES:
Tumor targeting pharmacokinetic parameters of iodine I 124 monoclonal antibody M5A | Days 0, 2, and 6 drawn at approximately 1 hour, 2 hour and 3-4 hours post-end of infusion
  Will be observed using standard imaging scans obtained pre-operatively and to assess if the antibody detects new liver metastases. Serum concentration data will be tabulated and descriptive statistics computed.
Percent of known liver lesions per standard staging scans identified on iodine I-124 (I-124) M5A imaging | Up to 1 year

SECONDARY OUTCOMES:
Surgical results (when available per standard of care surgery/pathology) on lesions negative on I-124 M5A but positive on standard scans | Up to 1 year
  percent of patients with pathological confirmation of liver metastases
Percent of patients with suspicious liver lesions identified on I-124 M5A but were not identified on standard imaging | Up to 1 year
Surgical pathology results (when available) on lesions positive on I-124 M5A but negative on standard imaging | Up to 1 year
  percent of patients with pathological confirmation of liver metastases
I-124 identification of extra-hepatic lesions (both previously noted or new) | Up to 1 year
  percent of patients with suspicious extra-hepatic lesions (both previously noted or new) identified on I-124 M5A but were not identified on standard imaging
Incidence of adverse events | Up to 14 days post infusion
  Will be graded according to Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. Safety data will be displayed and abnormal laboratory values reported. The frequency of adverse events will be tabulated by body system.

CONTACTS AND LOCATIONS:
Overall Officials: Savita V Dandapani, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States